CLINICAL TRIAL: NCT06042972
Title: Risk of Maternal Depression From 1 Year to 4 Years Postpartum in Yvelines
Acronym: DeTaPoP
Status: Recruiting | Type: Observational
Sponsor: Centre Médical Porte Verte (Other)
Responsible Party: Principal Investigator, Cyriane Courtois, Principal Investigator, Centre Médical Porte Verte
Other Study IDs: 2023-A01411-44
Record Dates: First submitted 2023-09-06; First posted 2023-09-21 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Post Partum Depression
Keywords: postpartum depression; depressive disorder; mental disorder; Edinburgh postnatal depression scale; EPDS; patient health questionnaire; PHQ2; pregnancy complications; puerperal disorders; moods disorders; maternity complications; behavioral symptoms; maternity; maternal distress; mental health; postnatal depression; social health; primary care
MeSH Terms: conditions — Depression, Postpartum; Depressive Disorder; Mental Disorders; Pregnancy Complications; Puerperal Disorders; Behavioral Symptoms; Psychological Well-Being | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire including Edinburgh postnatal depression scale, Patient Health Questionnaire 2 and background variables — Patients meeting the inclusion criteria will be recruited by health professionals who have agreed to participate in the study.
  Patients must fill out an anonymous self-questionnaire which will consist of 2 tests aimed to help diagnose postpartum depression, recommended in France by the Haute Autorité de Santé (HAS), and background variables.
  The self-questionnaire will be given back by the patient in a sealed envelope. Each questionnaire will only be filled out once per patient.

SUMMARY:
This observational study aims to estimate the prevalence of women from 1 to 4 years postpartum in Yvelines, who are suspected to suffer from postpartum depression, using the Edinburg Post natal Depression Scale (EPDS) and the Patient Heath Questionnaire 2 (PHQ2) and evaluate the factors that could be linked to it.

DETAILED DESCRIPTION:
The majority of studies and literature on maternal psychology focus on mothers of infants and newborns. The psychological experience of mothers with older children is still yet to be one of the subjects covered in the research on maternal psychology.

Postpartum depression characterizes itself in a depressive episode without psychotic characteristics, where symptoms appear in the year following delivery.

These symptoms reach their peak between 3 and 6 weeks postpartum. The diagnosis of postpartum depression is made by health professionals with the help of questionnaires such as the Edinburgh Postnatal Depression Scale (EPDS) or the Patient Health Questionnaire 2 (PHQ2).

According to the last national perinatal survey from Santé Publique France (Edition 2021), the rate of women having postpartum depression was estimated at 16.7%.

In France, the current psychological follow-up exam for women after giving birth includes a postnatal interview which is systematically offered between the 4th and the 8th week after delivery. It can be followed by another interview between the 10th and 14th week postpartum if judged necessary by the healthcare provider. It can also be offered by request.

Currently, there are no screening consultations for postpartum depression beyond the 14th week postpartum. Health care professionals are trained to be vigilant in the 1st year postpartum but not beyond this time frame.

A multicentric Australian study based on 1,507 women described the prevalence of maternal depression from early pregnancy to 4 years postpartum. It also covered the risk factors for depressive symptoms at 4 years postpartum.

The study concluded that maternal depression is more common at 4 years postpartum than at any time in the first 12 months postpartum. The prevalence of depressive symptoms at 4 years postpartum was 14.5% which was higher than at any time-point in the first 12 months post partum.

Currently, no French study focuses on the number of women suffering from maternal depression beyond 12 months postpartum.

This study aims to assess the prevalence of women 1 to 4 years postpartum who are suspected to have maternal depression and its linked factors.

Depression in one's lifetime can lead to negative consequences on a mother's psychological health and her quality of life, as well as her children's health.

The impact on children can include physical or mental developmental delay, regressed cognitive or language development, and general infant health issues.

Thus, if this study shows a significant risk for women to develop delayed maternal depression, extending a psychological follow-up exam of women beyond the 1st year postpartum could be necessary.

Moreover, screening and treating these women could limit the consequences on their children's development and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old
* Women from 1 year to 4 years postpartum or having children aged from 1 to 4 years old
* Patient gave their consent to participate in the study
* Patient lives in Yvelines
* Patient speaks and understands French
* Patient reads and writes in French

Exclusion Criteria:

* Patient suffered from postpartum depression in the 1st year after giving birth or is currently being treated for postpartum depression that started showing symptoms in the 1st year after giving birth.
* Patient is currently pregnant
* Patient gave birth less than 1 year prior or more than 4 years prior; or has a child who is less than one year old; or 5 or more years old
* Patient didn't give her consent to participate in the study
* Patient is under guardianship or judicial safeguard

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mothers of children aged from 1 year to 4 years living in Yvelines
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale and Patient Health Questionnaire 2 | Through study completion, an average of 10 months
  The primary outcome is positive if the Edinburgh Postnatal Depression Scale (EPDS) or the Patient Health Questionnaire 2 (PHQ2) are positive, meaning a score superior or equal to 10.5 for the EPDS or a score superior or equal to 3 for the PHQ2

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Porte Verte, Versailles, Île-de-France Region, France

REFERENCES:
- [Background] Woolhouse H, Gartland D, Mensah F, Brown SJ. Maternal depression from early pregnancy to 4 years postpartum in a prospective pregnancy cohort study: implications for primary health care. BJOG. 2015 Feb;122(3):312-21. doi: 10.1111/1471-0528.12837. Epub 2014 May 21. PMID 24844913
- [Background] Slomian J, Honvo G, Emonts P, Reginster JY, Bruyere O. Consequences of maternal postpartum depression: A systematic review of maternal and infant outcomes. Womens Health (Lond). 2019 Jan-Dec;15:1745506519844044. doi: 10.1177/1745506519844044. PMID 31035856
- [Background] Stein A, Pearson RM, Goodman SH, Rapa E, Rahman A, McCallum M, Howard LM, Pariante CM. Effects of perinatal mental disorders on the fetus and child. Lancet. 2014 Nov 15;384(9956):1800-19. doi: 10.1016/S0140-6736(14)61277-0. Epub 2014 Nov 14. PMID 25455250
- [Background] Depression and Suicide Screening Gregory Plemmons MD, MFA, in Adolescent Health Screening: an Update in the Age of Big Data, 2019
- [Background] Référentiel de psychiatrie. Collège national des universitaires en psychiatrie. Presses universitaires François Rabelais, 3ème édition, 2021
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Guedeney N, Fermanian J. Validation study of the French version of the Edinburgh Postnatal Depression Scale (EPDS): new results about use and psychometric properties. Eur Psychiatry. 1998;13(2):83-9. doi: 10.1016/S0924-9338(98)80023-0. PMID 19698604
- [Background] Murray L, Carothers AD. The validation of the Edinburgh Post-natal Depression Scale on a community sample. Br J Psychiatry. 1990 Aug;157:288-90. doi: 10.1192/bjp.157.2.288. PMID 2224383
- See also: Related Info — https://www.acog.org/clinical/clinical-guidance/committee-opinion/articles/2018/11/screening-for-perinatal-depression?utm_source=redirect&utm_medium=web&utm_campaign=otn
- See also: EPDS Français — http://www.perinatalservicesbc.ca/Documents/Resources/HealthPromotion/EPDS/EdinburghEPDSScale_French.pdf
- See also: PHQ2 — https://www.hiv.uw.edu/page/mental-health-screening/phq-2
- See also: Enquête Nationale Périnatale 2021 — https://www.santepubliquefrance.fr/les-actualites/2022/sante-publique-france-partenaire-de-la-6e-edition-de-l-enquete-nationale-perinatale
- See also: Related Info — https://www.msdmanuals.com/fr/professional/gyn%C3%A9cologie-et-obst%C3%A9trique/soins-du-post-partum-et-troubles-associ%C3%A9s/d%C3%A9pression-du-post-partum
- See also: Recommandations Haute Autorité de Santé dépression de l'adulte — https://www.has-sante.fr/upload/docs/application/pdf/2017-10/depression_adulte_recommandations_version_mel.pdf
- See also: Manuel de gynécologie et obstétrique: soins du post partum et troubles associés — https://www.msdmanuals.com/fr/professional/gynécologie-et-obstétrique/soins-du-post-partum-et-troubles-associés/dépression-du-post-partum